CLINICAL TRIAL: NCT07407140
Title: A Multicenter, Randomized, Controlled Trial of a Triple-Drug Regimen (Venetoclax, Azacitidine, Gilteritinib) Followed by Intensive Chemotherapy, Versus Standard Chemotherapy Plus Gilteritinib, in Fit Adults With Newly Diagnosed FLT3-Mutated Acute Myeloid Leukemia.
Brief Title: VAG Versus Standard Chemotherapy With FLT3 Inhibitor in Adult Patients With FLT3-Mutated AML
Acronym: VAG-3+7-G
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2026012
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: AML, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — gilteritinib; Azacitidine; venetoclax; Cytarabine; Daunorubicin; Idarubicin; Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VAG Induction (Experimental): Venetoclax (oral, dose ramp-up: 100 mg D1, 200 mg D2, 400 mg D3 onward), Azacitidine (75 mg/m²/day, D1-7), and Gilteritinib (120 mg daily) are administered as follows:
  Age <60 years: Venetoclax and Gilteritinib are given from D1-14. A bone marrow aspirate on D14 is required. If blasts are >5% with hypercellular marrow, both drugs may be extended to D21.
  Age ≥60 years: Venetoclax and Gilteritinib are given from D1-7. A bone marrow aspirate on D7 is required. If blasts are >5% with hypercellular marrow, both drugs may be extended to D14.
  Interventions: Drug: Gilteritinib + Azacitidine + Venetoclax; Drug: Re-induction Therapy; Drug: Consolidation Therapy; Drug: Maintenance Therapy
- Standard "3+7" plus gilteritinib induction (Active Comparator): Cytarabine (100 mg/m²/day continuous infusion, days 1-7) + Daunorubicin (60 mg/m²/day, days 1-3) OR Idarubicin (12 mg/m²/day, days 1-3)+ Gilteritinib (120mg, d8-21)
  Interventions: Drug: Cytarabine + Daunorubicin (or Idarubicin) + Gilteritinib; Drug: Re-induction Therapy; Drug: Consolidation Therapy; Drug: Maintenance Therapy

INTERVENTIONS:
Drug: Gilteritinib + Azacitidine + Venetoclax — Patients randomized to this arm receive the novel triplet combination as first-line induction therapy. Patients who achieve complete remission (CR) will receive one repeat cycle of the induction therapy.
  Arms: VAG Induction
Drug: Cytarabine + Daunorubicin (or Idarubicin) + Gilteritinib — Patients randomized to this arm receive the standard "3+7" intensive chemotherapy plus gilteritinib as the control regimen.
  Arms: Standard "3+7" plus gilteritinib induction
Drug: Re-induction Therapy — Gilteritinib: 80 mg daily, days 1-28.
  Azacitidine: 75 mg/m²/day, days 1-7.
  Venetoclax: Ramp-up: 100 mg (day 1), 200 mg (day 2), 400 mg daily (days 3-14).
  If Day 14 marrow blasts >5%, Venetoclax continues at 400 mg daily from days 14-21.
Drug: Consolidation Therapy — Applicable to: All patients achieving CRc (CR/CRh/CRi) following two cycles of induction in the experimental arm or one to two cycles in the control arm.
  Regimen: Intermediate-dose Cytarabine followed by Gilteritinib per group-specific criteria.
  Cytarabine (Both Arms):
  Age <60 years: 2 g/m² IV q12h, Days 1-3. Age ≥60 years: 1 g/m² IV q12h, Days 1-3.
  Gilteritinib Addition (120 mg oral, Days 4-17):
  Control Arm: Administered routinely in all patients. Experimental Arm: Added only if an FLT3 mutation is detectable by NGS-based MRD testing prior to the start of each consolidation cycle.
Drug: Maintenance Therapy — Applicable to: All patients who have completed consolidation therapy.
  Experimental Arm: Adjusted-dose VA regimen for 6 cycles.
  Azacitidine: 75 mg/m²/day, Days 1-7.
  Venetoclax: 400 mg daily, Days 1-7.
  Control Arm: Gilteritinib monotherapy for up to 1 year.
  Gilteritinib: 120 mg daily, Days 1-365.

SUMMARY:
This prospective, multicenter, randomized, open-label, controlled trial compares the efficacy and safety of two induction regimens in adults with newly diagnosed, FLT3-mutated AML who are eligible for intensive chemotherapy. Approximately 300 patients aged ≥14 years will be randomized 1:1 to receive either induction with the VAG regimen (Venetoclax, Azacitidine, and Gilteritinib) or with the standard "3+7" regimen (Cytarabine plus Daunorubicin/Idarubicin) with Gilteritinib. Patients in the experimental arm achieving complete remission will receive one additional cycle of the VAG regimen.

Those who do not achieve remission after the first induction cycle will receive one cycle of VAG as re-induction, irrespective of initial assignment. Patients who enter remission will proceed to consolidation with three cycles of intermediate-dose cytarabine. During consolidation, Gilteritinib will be continuously given in the control arm, while in the experimental arm, it will be added only if FLT3 mutation is detected by NGS-based MRD testing prior to consolidation. Subsequently, maintenance therapy will be administered: the experimental arm will receive 6 cycles of VA (Venetoclax and Azacitidine), and the control arm will receive Gilteritinib for up to one year. Allogeneic hematopoietic stem cell transplantation is permitted for eligible intermediate- or high-risk patients in remission. The primary endpoint is Overall Survival (OS).

DETAILED DESCRIPTION:
FLT3 mutations confer poor prognosis in AML, and resistance remains a challenge despite current FLT3 inhibitor-based therapies. Preclinical and early clinical data support the potent efficacy of the triple combination of Venetoclax, Azacitidine, and Gilteritinib (VAG). This study aims to determine if VAG induction is superior to standard "3+7" chemotherapy plus gilteritinib in fit, FLT3-mutated AML patients. The trial includes a VAG salvage strategy for non-responders and a stratified post-remission pathway for all responders.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AML (excluding CBF-AML and APL) or MDS/AML (with 10%-20% marrow blasts) per WHO 2022 or ICC criteria
* Documented FLT3-ITD or FLT3-TKD mutation by PCR or NGS
* Age ≥14 and <75 years
* Eligible for intensive chemotherapy
* ECOG performance status 0-2
* Adequate organ function (liver, kidney, cardiac)
* Written informed consent

Exclusion Criteria:

* Acute promyelocytic leukemia with PML-RARA
* Core-binding factor AML (RUNX1-RUNX1T1 or CBFB-MYH11)
* BCR-ABL positive AML
* Prior induction chemotherapy for AML (hydroxyurea allowed)
* Concurrent active malignancy requiring therapy
* Active/symptomatic cardiac disease
* Severe uncontrolled infection
* Any condition deemed unsuitable by the investigator

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From randomization until death from any cause, assessed up to 3 years

SECONDARY OUTCOMES:
Composite Complete Remission Rate | After induction therapy (approximately 4-8 weeks)
Measurable residual disease-negative CRc rate by flow cytometry | At the time of achieving CRc
  Measurable residual disease-negative CRc rate by flow cytometry after every courses therapy
Measurable residual disease-negative CRc rate by NGS for FLT3-ITD | At the time of achieving CRc
  Measurable residual disease-negative CRc rate by NGS for FLT3-ITD after every courses therapy
Event-Free Survival (EFS) | From randomization until treatment failure, relapse after CRc, death from any cause, or last follow-up, assessed up to 3 years
Relapse-Free Survival (RFS) | From achievement of CRc until relapse, death, or last follow-up, assessed up to 3 years
30-day and 60-day mortality | 30 and 60 days after start of induction therapy